CLINICAL TRIAL: NCT04402112
Title: Efficacy and Safety of Pitavastatin in a Real-wOrld Setting: Observational Study Evaluating saFety in Patient With Pitavastatin for Lipid Lowering Therapy in Korea
Brief Title: Efficacy and Safety of Pitavastatin in a Real-world Setting
Acronym: PROOF
Status: Completed | Type: Observational
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: JWP-PTV-712
Record Dates: First submitted 2020-04-27; First posted 2020-05-26 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Hypercholesterolemia
Keywords: Pitavastatin; LIVALO; Safety data; South Korea; Large-scale prospective trial
MeSH Terms: conditions — Hypercholesterolemia | interventions — pitavastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Pitavastatin — 1mg, 2mg, or 4mg, Once a day, at least 8 weeks
  Other Names: LIVALO

SUMMARY:
The prospective, observational, non-comparative trial in South Korea was designed to evaluate the efficacy and safety of pitavastatin (Livalo) in clinical practice in 28,343 patients.

DETAILED DESCRIPTION:
This study was conducted in 893 facilities in Korea from 2 Apr 2012 to 1 Apr 2017. This study was designed to administer 1mg, 2mg, or 4mg pitavastatin to patients with hyperlipidemia at the age of 20 or older for at least 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of statin treatment who are taking or are planning to take Livalo tablets, or who are taking other statins or are planning to change to Livalo tablets.

Exclusion Criteria:

* Patients with hypersensitivity to pitavastatin
* Patients with active liver disease or untranslated transaminase levels Patients with a constant rise in
* Patients with severe liver failure or biliary obstruction and patients with cholestasis
* Patients who are receiving cyclosporine
* Myopathy patients
* Pregnant women or women of childbearing age and lactating women
* Children
* Patients with genetic problems, such as galactose intolerance, Lapp lactose deficiency or glucose-galactose
* Patients deemed inappropriate by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving Livalo tablets in clinical practice in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 28343 (Actual)
Dates: Start 2012-04-02 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v4.0 | At 8 weeks after administration of pitavastatin
  Incidence of musculoskeletal-related adverse events and rhabdomyolysis

SECONDARY OUTCOMES:
Overall symptom satisfaction evaluation | At 8 weeks after administration of pitavastatin
  The investigating physician selects one of the followings according to medical judgment: Improvement, constant, exacerbation
Change in serum lipid profile before and after administration of pitavastatin | At screening and after 8 weeks
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglyceride

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Rae Kim, MD,PhD, Principal Investigator — The Catholic University of Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jeong IK, Kim SR. Efficacy and Safety of Pitavastatin in a Real-World Setting: Observational Study Evaluating SaFety in Patient Treated with Pitavastatin in Korea (PROOF Study). Endocrinol Metab (Seoul). 2020 Dec;35(4):882-891. doi: 10.3803/EnM.2020.723. Epub 2020 Dec 2. PMID 33261312